CLINICAL TRIAL: NCT03490396
Title: An Adaptive Design, Single-Blind, Randomized, Controlled Study Investigating Polyvinylpyrrolidone (PVP) and Sodium Hyaluronate-Containing Oral Gel (Gelclair®) in Comparison to Viscous Lidocaine, Diphenhydramine, and Aluminum-magnesium Hydroxide/Simethicone Antacid Suspension Mouthwash ("Magic Mouthwash") for the Management of Oral Mucositis Associated With High Dose Chemotherapy and Methotrexate in Allogeneic Stem Cell Transplant Recipients
Brief Title: Gelclair at Conditioning or After Oral Mucositis Diagnosed vs. Magic Mouth Wash in Stem Cell Transplant Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Midatech Pharma US Inc. (Industry)
Collaborators: PharPoint Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GEL-401
Record Dates: First submitted 2018-03-14; First posted 2018-04-06 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; Stomatitis; Myeloablative
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: The initial design is a prospective, randomized, single-blind (evaluator), parallel, three arm, controlled clinical study.
Who Masked: Outcomes Assessor
Masking Description: OM grading via the WHO oral toxicity grading scale will be performed by the trained blinded evaluator at least 3X/week (e.g., M, W and F), with ≤ 48h (±24h) in between each assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm 1 (Gelclair at time of conditioning) (Experimental): All subjects in study Arm 1 will receive GEL starting on the first day of conditioning.
  Interventions: Device: Gelclair
- Arm 2 (Gelclair when OM diagnosed) (Active Comparator): Subjects in Arm 2 will be observed from initiation of conditioning to Day +14. If subjects develop G1 or G2 OM via WHO OM scale during this period, they will at that time be randomized to immediately receive GEL.
  Interventions: Device: Gelclair
- Arm 3 (MMW when OM diagnosed) (Active Comparator): Subjects in Arm 2 will be observed from initiation of conditioning to Day +14. If subjects develop G1 or G2 OM via WHO OM scale during this period, they will at that time be randomized to immediately receive MMW.
  Interventions: Combination Product: First® Mouthwash BLM

INTERVENTIONS:
Device: Gelclair — Polyvinylpyrrolidone (PVP) and Sodium Hyaluronate-Containing Oral Gel
  Other Names: Gelclair Bioadherent Oral Gel
  Arms: Arm 1 (Gelclair at time of conditioning); Arm 2 (Gelclair when OM diagnosed)
Combination Product: First® Mouthwash BLM — Viscous Lidocaine, Diphenhydramine, and Aluminum-magnesium Hydroxide/Simethicone Antacid Suspension Mouthwash
  Other Names: Magic Mouth Wash
  Arms: Arm 3 (MMW when OM diagnosed)

SUMMARY:
Patients receiving high-dose chemotherapy/conditioning prior to stem cell transplantation (SCT) are at high risk for developing painful lesions in the oral cavity, known as oral mucositis (OM).

In this high risk adult population, the study objectives are to investigate the efficacy and tolerability of Gelclair® (GEL; an FDA cleared medical device indicated for the management of painful oral lesions) and ideal timing of initiation of therapy (at the time of conditioning or after mild OM is diagnosed) for the management of oral mucositis (OM), relative to a commercially available compounded mouth wash (First® Mouthwash BLM "Magic Mouth Wash"; MMW) initiated after mild OM is diagnosed. The study may be adapted based on an interim analysis and recommendations of the interim data review committee.

DETAILED DESCRIPTION:
Adult patients at high risk for developing OM receiving one of the following myeloablative (MA) pre-transplant conditioning regimens prior to allogeneic transplant along with methotrexate (MTX) as part of graft vs. host disease (GVHD) prophylaxis meeting all other eligibility criteria will be enrolled:

* FluBu based regimens: either fludarabine: 30 mg/m^2 x 4 days and busulfan 0.8 mg/kg IV q6h x 4 days; both given daily starting at day -4 OR fludarabine: 40 mg/m^2 and busulfan: 3.2 mg/kg both given daily on days -6 through -3.
* Bu/Cy: busulfan, 0.8 mg/kg IV q6h x 4 days (-7 through -4); cyclophosphamide: 60 mg/kg IV once on days -3 and -2
* Cy/TBI: Cyclophosphamide, 60 mg/kg IV given twice between days -3 and -1 and TBI fractionated (generally over 3 days) for a total of 12Gy

GVHD Prophylaxis:

• Regimens including methotrexate (MTX; 15 mg/m^2 planned to be given on days 1, 3, 6 and 11); addition of other agents given along with MTX (e.g., tacrolimus, sirolimus) is acceptable.

Duration of treatment:

* Arm 1: GEL treatment a minimum of 4x/day initiated from 1st day of conditioning through OM resolution (G0), up to a maximum of 20d.
* Arms 2 (GEL) and 3 (MMW): Treatment a minimum of 4x/day initiated when G1 or G2 OM diagnosed during observation period (through Day +14 relative to stem cell infusion) through OM resolution (G0), up to a maximum of 20d.

ELIGIBILITY:
Inclusion Criteria:

* Be age ≥ 18 years old.
* Have Karnofsky performance status score ≥ 70.
* Be scheduled to receive one of 3 myeloablative conditioning regimens (defined in population) followed by allogeneic SCT for hematological malignancy.
* Have anticipated in-patient status for 14 to 20 days from the time of transplant.
* Be willing and capable of swishing/gargling oral gel/solution as required per protocol.
* Be willing and capable of completing the assessments and adhering to protocol requirements.
* Be willing and able to provide written informed consent.

To be randomized to begin treatment, subjects randomized to Arms 2 or 3 must also meet the following criterion:

-Be diagnosed with G1 or G2 OM via WHO OM scale during observation period from conditioning to Day +14.

Exclusion Criteria:

* Subjects receiving pre-transplant conditioning/GVHD prophylaxis regimens other than those defined, herein.
* Use of topical or systemic agents/treatments for OM within 2 weeks of treatment day 1.
* Evidence of uncontrolled infection (oral/oropharyngeal or systemic), including oral herpes or unexplained febrile illness (≥ 99.5F /37.5C) requiring systemic anti-infectives, within 7d of treatment Day 1.
* Subjects with active oral lesions or other mouth/throat soreness within 7d of study randomization.
* Any other criteria, in the opinion of the investigator that would make the subject unsuitable for study participation.

For subjects randomized to Treatment Arms 2 or 3 during observation period:

-OM ≥ G3 diagnosed prior to initiating randomized treatment during observation period (conditioning through Day +14; i.e., missed treatment window).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence/occurrence of any grade Oral Mucositis | Initial study period (initiation of conditioning through day +14 post-transplant)
  Incidence/develop of any grade of OM as assessed via WHO OM grading scale (Grades possible: 1-4)
Area under the curve in mouth and throat soreness (MTS) | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)

SECONDARY OUTCOMES:
Time to onset of any grade OM | Initial study period (initiation of conditioning through day +14 post-transplant)
  WHO Grades 1-4
Duration of any grade OM | Study period (initiation of conditioning through day +28 post-transplant)
  WHO Grades 1-4
Severity of OM | Study period (initiation of conditioning through day +28 post-transplant)
  WHO Grades 1-4
Incidence of severe OM | Study period (initiation of conditioning through day +28 post-transplant)
  WHO Grades 3-4
Time to onset of severe OM | Study period (initiation of conditioning through day +28 post-transplant)
  WHO Grades 3-4
Duration of severe OM | Study period (initiation of conditioning through day +28 post-transplant)
  WHO Grades 3-4
Magnitude of OM-related pain control | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  Based on subject grading of mouth and throat soreness (VAS 0 (no pain) to 10 (max pain possible)) prior to each randomized/rescue OM treatment.
Duration of pain control | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  Based on time at a given mouth and throat soreness level and/or need for rescue treatment to control mouth and throat soreness.
Opiate and other background pain medication use | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)

OTHER OUTCOMES:
Weight change over study treatment period | Study period (initiation of conditioning through day +28 post-transplant)
Incidence of treatment-emergent infection | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  e.g., bacteremia/febrile neutropenia, including oral infections (e.g., thrush).
Duration of treatment-emergent infections | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  e.g., bacteremia/febrile neutropenia, including oral infections (e.g., thrush).
Use of anti-infectives for treatment-emergent infections | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  Exploratory Endpoint
Duration of anti-infective use for treatment-emergent infections | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
Dose level of anti-infectives for treatment-emergent infections | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
Days of hospitalization post-SCT | Study period (initiation of conditioning through day +28 post-transplant)
Incidence of need for a modified diet | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  For example, soft, liquid, TPN
Duration of need for a modified diet | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
  For example, soft, liquid, TPN
Treatment Compliance with randomized OM treatment | Study period (initiation of conditioning through day +28 post-transplant)
  Assessed by determining the number of randomized treatments actually taken relative to the number of treatments required (i.e., treatment compliance)
Use of rescue treatments other than randomized agent for managing OM | While OM ongoing during study period (initiation of conditioning through day +28 post-transplant)
Incidence of treatment-emergent xerostomia ≥ G2 | Study period (initiation of conditioning through day +28 post-transplant)
Duration of treatment-emergent xerostomia ≥ G2 | Study period (initiation of conditioning through day +28 post-transplant)
Use of treatments/medications to manage xerostomia | Study period (initiation of conditioning through day +28 post-transplant)
Duration of use for treatments/medications to manage xerostomia | Study period (initiation of conditioning through day +28 post-transplant)
Impact of OM on activities of daily living | Study period (initiation of conditioning through day +28 post-transplant)
  Via validated oral mucositis daily questionnaire (OMDQ)
Diarrhea associated with OM | Study period (initiation of conditioning through day +28 post-transplant)
  Via validated oral mucositis daily questionnaire (OMDQ)
Exploratory Safety/Tolerability of GEL and MMW | Study period (initiation of conditioning through day +28 post-transplant)
  Assessed by treatment-emergent and related adverse events/serious adverse events/unanticipated adverse device effects and subject reported tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Delmedico, PhD, Study Director — Midatech Pharma US Inc.
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital/Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gelclair Website (Study Agent) — http://www.gelclair.com/